CLINICAL TRIAL: NCT03939988
Title: Evaluation of the Use of Photobiomodulation After the Installation of Elastometric Separators - Randomized Controlled Clinical Trial.
Brief Title: Evaluation of the Use of Photobiomodulation After the Installation of Elastometric Separators
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Silvana
Record Dates: First submitted 2019-05-04; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Orthodontic Appliance Complication
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Masking Description: In the Placebo group, participants will receive the simulated application with the laser set off, only using the beep to play the application. Therefore, they not know to which group they belong.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): In this study, immediately after the installation of the separators, the subjects of the experimental group will be submitted to photobiomodulation. The laser will be infrared, in continuous mode with wavelength of 808 nm. The tip will be positioned perpendicularly in the mucosa, without exerting pressure. At each point 2J of energy will be irradiated for 20 seconds, totaling 12J per tooth, 6J on the buccal side and 6J of the lingual side of the teeth.
  Interventions: Radiation: Photobiomodulation
- Placebo group (Placebo Comparator): In the placebo group, the same procedures will be made, but the laser will be switched off.
  Interventions: Radiation: Placebo photobiomodulation

INTERVENTIONS:
Radiation: Photobiomodulation — Immediately after the installation of the separators, the subjects will be submitted to photobiomodulation. The laser will be infrared, in continuous mode with wavelength of 808 nm. The tip will be positioned perpendicularly in the mucosa, without exerting pressure. At each point 2J of energy will be irradiated for 20 seconds, totaling 12J per tooth, 6J on the buccal side and 6J of the lingual side of the teeth.
  Arms: Experimental group
Radiation: Placebo photobiomodulation — In the placebo group, the same procedures will be made, but the laser will be turned off.
  Arms: Placebo group

SUMMARY:
The greatest dropout rate of orthodontic treatments is pain, from the installation of the elastomeric separators, to the exchange of wires and accessories. This process that presents both physiological and psychological responses negatively affects patients' quality of life due to the difficulty of chewing and biting. The sample will be comprised of individuals who will receive elastomeric spacers on the mesial and distal surfaces of the upper first molars, randomized into two groups, the group being irradiated with the low intensity laser, called the experimental group, and the placebo group, simulated laser. In the installation of the tabs, the experimental group will receive a single application in the mesial and distal cervical portion and in the apical third of the molars. The energy delivered at each point will be 2J, per vestibular and lingual, 6 points, totaling 12 J of energy per tooth. To evaluate the perception of pain we will use the Visual Analogue Scale (EVA) after 1h, for all groups. The gingival pockets cytokines will be collected with an absorbent paper cone for 30 seconds on both groups and compared between them by ELISA. It is expected that patients in the irradiated group will have lower pain perception and less cytokines than in the placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Clinical conditions of normality;
* Healthy periodontium;
* Healthy molars;
* Presence of interproximal contacts between the second molar and premolar;
* Permanent dentition phase;
* Who have not been taking anti-inflammatory drugs or analgesics for 4 days.

Exclusion Criteria:

* Systemic diseases that routinely use medications;
* Patients with periodontal disease;
* Patients who remove the tabs or who do not respond to the questionnaire;
* Papers contaminated with blood or saliva will be excluded for cytokine analysis.

Ages: 12 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (pain measurement) | Immediately after treatment.
  After an hour of installation of the separators, patients will respond to pain perception, being instructed to quantify their level of discomfort by measuring the VAS. The scale was converted into 11 points, 0 to 10, where 0 refers to the absence of pain and 10 levels of intolerable pain.

SECONDARY OUTCOMES:
Change in IL-8 cytokine | Baseline and immediately after treatment.
  We will insert absorbent tissue cones at the sampling sites (gingival pockets), before and one hour after the insertion of the separators. The levels of cytokines will be analyzed by the ELISA interleukin kits method, strictly following the manufacturer's instructions, by the same examiner.

REFERENCES:
- [Derived] Ortega SM, Goncalves MLL, da Silva T, Horliana ACRT, Motta LJ, Altavista OM, Olivan SR, Santos AECGD, Martimbianco ALC, Mesquita-Ferrari RA, Fernandes KPS, Bussadori SK. Evaluation of the use of photobiomodulation following the placement of elastomeric separators: Protocol for a randomized controlled clinical trial. Medicine (Baltimore). 2019 Oct;98(43):e17325. doi: 10.1097/MD.0000000000017325. PMID 31651838